CLINICAL TRIAL: NCT00189254
Title: A Follow-up Study to Evaluate Actinic Keratosis Recurrence Rates One Year After Completion of the 1487-IMIQ Study
Brief Title: A Study to Follow up Recurrence Rates of Actinic Keratoses One Year After Completion of Study 1487-IMIQ
Status: Completed | Type: Observational
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: 1524-IMIQ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2015-04

CONDITIONS: Actinic Keratoses
Keywords: 1 year follow up
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Imiquimod 5% cream: No investigational treatments were given during this study.
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — No defined treatments were given during this study.

SUMMARY:
The purpose of the study is to obtain recurrence rates and long-term safety data for patients who had been treating actinic keratoses on the face and scalp with 5 % Imiquimod Cream in a previous study.

ELIGIBILITY:
Inclusion Criteria:

* 100% clearance of Actinic Keratosis (AK) lesions in the 1487 IMIQ study

Exclusion Criteria:

* used any treatments in the previous treatment area within 24 hours prior to the follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At least 18 years old. Females of childbearing potential, with a negative urine pregnancy test, must have been willing to use a medically acceptable method of contraception during the treatment.
Sampling Method: Probability Sample
Enrollment: 72
Dates: Start 2005-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Efficacy | one year after completion of study 1487-Imiq
  Efficacy was evaluated by counting AK lesions in the previous treatment area. Subjects at the 1-year follow-up visit with recurrence of lesion(s).
Safety | one year after completion of study 1487-Imiq
  Safety was evaluated by assessing the area of previous treatment for LSRs and skin quality
Adverse Events | one year after completion of study 1487-Imiq
  AEs considered by investigator to be possibly or probably related to the 1487-Imiq study medication were documented and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Study Coordinator, Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau